CLINICAL TRIAL: NCT02552576
Title: An Open-label, Multi-centre Post-marketing Study to Assess the Efficacy and Safety of Voncento® in Subjects With Von Willebrand Disease
Brief Title: Study of Voncento® in Subjects With Von Willebrand Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-BIO-12-83; 2013-003305-25 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voncento (Experimental): The frequency and dose of Voncento administration will be determined by the investigator using the information included in the Voncento Summary of product characteristics (SmPC)
  Interventions: Biological: Voncento

INTERVENTIONS:
Biological: Voncento — Human coagulation VWF / coagulation factor VIII (FVIII) complex concentrate

SUMMARY:
This is a multi-centre, open-label, single-arm, phase 4, post-marketing study to further investigate the efficacy and safety of Voncento in subjects with Von Willebrand Disease (VWD) in whom treatment with a Von Willebrand Factor (VWF) product is required as on-demand therapy, for prophylactic therapy, or during surgery. Subjects will be treated with Voncento either as an on-demand regimen (eg, to treat a non-surgical spontaneous or traumatic bleeding event) or prevention regimen (eg, to prevent an anticipated bleeding event) at a dose prescribed by the Investigator in accordance with the Voncento Summary of Product Characteristics (SmPC), or with a prophylaxis regimen (regular treatment with Voncento at a frequency of 1-3 times per week). Voncento will also be given to prevent and treat any surgical bleeding events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe type 1, 2A, or 3 VWD where Von Willebrand Factor: Ristocetin Cofactor (VWF:RCo) is <20% at screening
* Desmopressin acetate treatment is ineffective, contraindicated, or not available for subject (type 3 VWD subjects only).
* Evidence of vaccination against hepatitis A and B or presence of antibodies against hepatitis A and B due to either a previous infection or prior immunization.
* Written informed consent given.
* Require a VWF product to control a non-surgical bleeding (NSB) event or for ongoing prophylactic therapy.

Exclusion Criteria:

* Known history or suspicion of having VWF or FVIII inhibitors
* Acute or chronic medical condition, other than VWD, which may affect the conduct of the study
* Known or suspected hypersensitivity or previous evidence of severe side effects to Voncento, VWF / FVIII concentrates, or human albumin.
* Participated in another interventional clinical study within 30 days before the first administration of Voncento or at any time during the study.
* Females who are pregnant, breast-feeding or who have a positive pregnancy test at screening
* Alcohol, drug, or medication abuse within 1 year before the study.
* Currently receiving a therapy not permitted during the study.
* Previous participation in a Voncento / Biostate study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Haemostatic efficacy - NSB event | Assessed daily by the subject until the bleed stops, for the duration of the subject's participation in the study (approximately 12 months). Each bleeding event is also to be assessed retrospectively by the Investigator.
  Subject's and investigator's assessment of haemostatic efficacy of Voncento in its usage for a non-surgical bleeding (NSB) event. Assessments of haemostatic efficacy will be based on a 4-point ordinal scale of Excellent, Good, Moderate or None.
Number of infusions - NSB event | For the duration of the subject's participation in the study (approximately 12 months).
  Number of infusions of Voncento required to treat an NSB event.
Total dose of Voncento - NSB event | For the duration of the subject's participation in the study (approximately 12 months).
  Total dose of Voncento (in international units of Von Willebrand Factor: Ristocetin Cofactor) required to treat an NSB event.
Number of NSB events per month | From Day 1 until final study visit, approximately 12 months.
Annual bleeding rate | For the duration of the subject's participation in the study (approximately 12 months).
  The number of bleeding events per year

SECONDARY OUTCOMES:
Assessment of blood loss during a surgical procedure | During surgery, for any surgical procedure during the subject's participation in the study (approximately 12 months).
Haemostatic efficacy - surgical event | Assessed during and after surgery until the bleeding stops, for any surgical procedure during the subject's participation in the study (approximately 12 months).
  Investigator's or surgeon's assessment of haemostatic efficacy of Voncento in its usage for a surgical bleeding event. Assessments of haemostatic efficacy will be based on a 4-point ordinal scale of Excellent, Good, Moderate or None.
Number of infusions - surgical bleeding event | For the duration of the subject's participation in the study (approximately 12 months).
  Number of infusions of Voncento required to treat a surgical bleeding event.
Total dose of Voncento - surgical bleeding event | For the duration of the subject's participation in the study (approximately 12 months).
  Total dose of Voncento (in international units of Von Willebrand Factor: Ristocetin Cofactor) required to treat a surgical bleeding event.
Overall adverse events | From Day 1 until the final study visit for each subject (approximately 12 months)
  Overall number of subjects with: adverse events (AEs), serious AEs, AEs related to Voncento administration, and adverse events of special interest.
Number of subjects with VWF or FVIII inhibitors | At screening, Day 1 and approximately Months 3, 6, 9 and 12, for each subject.
Haemostatic efficacy - prophylaxis | Approximately every month (subject assessment) and every 3 months (Investigator assessment) for the duration of the subject's participation in the study (approximately 12 months).
  Subject's and investigator's assessment of haemostatic efficacy of Voncento as prophylaxis therapy. Assessments of haemostatic efficacy will be based on a grading scale with outcomes of excellent, good, moderate, none.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (12):
- Study Site, Vienna, Austria
- Germany (2):
  - Study Site, Duisburg
  - Study Site, Frankfurt
- Study Site, Athens, Greece
- Poland (3):
  - Study Site, Krakow
  - Study Site, Rzeszów
  - Study Site, Wroclaw
- United Kingdom (5):
  - Study Site 14, London
  - Study Site 40, London
  - Study Site 42, London
  - Study Site 47, London
  - Study Site 8, London